CLINICAL TRIAL: NCT01164046
Title: Long-term Treatment for Cancer Patients With Deep Venous Thrombosis or Pulmonary Embolism
Acronym: Longheva
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to slow inclusion of patients
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Pieter W. Kamphuisen, MD PhD, Prof, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT nr: 2009-015336-15; Protocol nr: 29462 (Other: CCMO The Netherlands)
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Venous Thromboembolism; Neoplasms
Keywords: anticoagulants; Heparin, Low-Molecular-Weight; 4-Hydroxycoumarins; recurrent venous thrombosis
MeSH Terms: conditions — Venous Thromboembolism; Neoplasms; Venous Thrombosis | interventions — Heparin, Low-Molecular-Weight; Nadroparin; Enoxaparin; Tinzaparin; bemiparin; reviparin; Dalteparin; certoparin; acarboxyprothrombin; Phenprocoumon; Acenocoumarol; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin K antagonists (Active Comparator)
  Interventions: Drug: vitamin K antagonists
- Low molecular weight heparin (Active Comparator)
  Interventions: Drug: low molecular weight heparin

INTERVENTIONS:
Drug: low molecular weight heparin — weight adjusted dose of low molecular weight heparin, any type allowed if approved, 65-75% of full therapeutic dose
  Other Names: nadroparin; enoxaparin; tinzaparin; bemiparin; reviparin; dalteparin; certoparin
  Arms: Low molecular weight heparin
Drug: vitamin K antagonists — Target INR between 2-3. Any type allowed, if approved for use in that country.
  Other Names: phenprocoumon; acenocoumarol; warfarin
  Arms: vitamin K antagonists

SUMMARY:
Background

Patients with cancer and a first deep venous thrombosis of the leg or pulmonary embolism (venous thromboembolism, VTE) are generally treated with low molecular weight heparin (LMWH)injections for 6 months, since this treatment is associated with a reduced incidence of recurrent VTE compared to vitamin K antagonists (VKA). It is recommended that patients with active malignancy (metastatic cancer and/or ongoing cancer treatment)continue anticoagulant treatment. However, it is unknown whether LMWH is still superior compared to VKA for the long-term anticoagulant treatment.

Aim

The aim of this study is to evaluate whether low-molecular-weight heparin more effectively reduces recurrent VTE compared to vitamin K antagonists in patients with cancer who have already completed 6 to 12 months of anticoagulant treatment because of deep venous thrombosis of the leg or pulmonary embolism.

Hypothesis

The investigators hypothesize that LMWH is more effective compared to VKA in the long-term treatment of VTE in cancer patients who have already been treated for 6-12 months with anticoagulants.

Design

This is a multicenter, multinational, randomized, open label trial.

Patients

Patients with a malignancy (all types, solid and hematological) who have received 6-12 months of anticoagulation for VTE and have an indication for continuing anticoagulation, will be randomly assigned to six additional months of LMWH or VKA. LMWH will be administered in a weight-adjusted scheme, with 65-75% of therapeutic doses. All types of LMWH and VKA are allowed, as long as weight adjusted dosing is possible for LMWH. The target INR will be 2.0-3.0. The primary efficacy outcome is symptomatic recurrent VTE, i.e. deep vein thrombosis and pulmonary embolism. The primary safety outcome is major bleeding.

Sample size

A total of 65 to 87 recurrent VTE events are needed to show a 50% reduction with LMWH as compared to VKA (type I error 0.05, two-sided, power respectively 80 and 90%). To observe 75 events, with a 10% event rate per half year in the VKA arm and 5% in the LMWH arm a total of 1000 patients will need to be included.

Organisation

Outcomes will be adjudicated by a central adjudication committee. A steering committee will be formed, preferably consisting of one member of every participating center. An electronic case report form will be used for data collection. Also, an electronic trial master file will be used.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE), including deep venous thrombosis (DVT) and pulmonary embolism (PE), represents a major cause of morbidity and mortality in cancer patients. 1 The risk of VTE is increased several-fold in patients with cancer with incidences ranging between 4% and 20%. 2 Treatment of VTE aims at preventing recurrent events, including potentially fatal PE, which in turn could reduce the morbidity, use of health care resources and, above all, mortality for cancer patients.

Standard treatment for VTE consists of an initial course of heparin followed by vitamin K antagonists (VKAs) with doses adjusted to maintain an international normalized ratio (INR) between 2.0 and 3.0. Several unique aspects related to the cancer itself and its management make VKA therapy more complex than in non cancer patients. Chemotherapy induced thrombocytopenia and invasive procedures, for instance, may require a temporary interruption of anticoagulant therapy and a prompt reversal of the anticoagulant effect. On the other side, poor nutrition, concomitant medications, and impaired liver function can cause unpredictable changes in the dose response of VKAs. In addition, VKAs seem less effective and safe in cancer patients who experience a 3-fold higher risk of VTE recurrence and a 3-fold higher risk of bleeding during anticoagulation compared to patients without cancer. 3-5 Most bleeding and thrombotic complications occur with anticoagulant parameters within the therapeutic range. Therefore, more aggressive anticoagulant therapy would have the potential to reduce the risk of recurrent VTE, but at the price of an increase in bleeding.

Recently, randomized clinical trials and prospective cohort studies in cancer patients with acute VTE have shown that low-molecular-weight heparin (LMWH) may be more effective in preventing VTE recurrences at a comparable bleeding risk as compared to VKA's. 6-9 In addition, LMWH offer the advantages of being easier to administer, more flexible, and not influenced by nutrition problems or liver impairment.

In the CLOT (Randomized Comparison of Low-Molecular-Weight Heparin Versus Oral Anticoagulant Therapy for the Prevention of Recurrent Venous Thromboembolism in Patients with Cancer) study, cancer patients with acute, symptomatic proximal DVT, PE, or both, were randomly assigned to receive dalteparin (200 IU/kg of body weight subcutaneously once daily for 5 to 7 days) followed by a coumarin derivative for 6 months, or dalteparin alone for 6 months (200 IU/kg of body weight once daily for 1 month followed by 150 IU/kg body weight once daily for 5 months). During the 6-month study period, 27 of 336 patients (9%) in the dalteparin group had symptomatic, objectively documented recurrent VTE as compared to 53 of 336 patients (17%) in the VKAs group, hazard ratio 0.48 (95% CI: 0.30, 0.77, p=0.002). There was no statistically significant difference in major bleeding (6% versus 4%, p=0.27) nor in any bleeding (14% and 19%, respectively, p=0.09) between the two study groups. 6 In a randomized, open-label multicenter trial, subcutaneous enoxaparin sodium (1.5 mg/kg once daily) was compared with warfarin given for 3 months in 146 cancer patients with VTE. 7 Fifteen (21.1%) of the 71 assessable patients assigned to receive warfarin had one major bleeding or a recurrent VTE within 3 months compared with seven patients (10.5%) of the 67 assessable patients assigned to receive enoxaparin (p=0.09). There were six deaths as a result of hemorrhage in the warfarin group compared with none in the enoxaparin group.

In a RCT of 122 cancer patients with acute symptomatic VTE, no significant differences in major and minor bleeding rates were observed between patients assigned to subcutaneous enoxaparin given for up to 180 days and those receiving enoxaparin followed by warfarin. 8 In the LITE (Longitudinal Investigation of Thromboembolism Etiology) study, cancer patients with acute symptomatic proximal DVT were randomized to intravenous UFH followed by VKAs for 3 months or tinzaparin (175 U/kg once daily) alone for 3 months. During the 1-year observational period, recurrent VTE occurred in 16 of 100 (16%) patients assigned to UFH-VKAs compared with 7 of 100 cancer patients (7%) treated with tinzaparin. 9 The American Society of Clinical Oncology and the American College of Chest Physicians guidelines advice LMWH for acute and long-term treatment in cancer patients with acute VTE. 10-11 The US Food and Drug Administration has recently approved dalteparin sodium for long-term treatment of symptomatic VTE in cancer patients. 12 Long-term anticoagulant therapy with VKAs is suggested when LMWH is not available.

After 6 months of LMWH, indefinite anticoagulant therapy is suggested for patients with active cancer, such as those with metastases or receiving chemotherapy. These patients are considered to be at a greater risk for recurrent VTE. For most patients, this means lifelong anticoagulation. The relative benefits and risks of continuing LMWH beyond 6 months versus switching to oral VKAs, remains a clinical judgment in the individual patient. Some experts in the field recommend VKAs in patients with less advanced disease. 13 The risks of long-term LMWH therapy include bleeding, heparin-induced thrombocytopenia and osteoporosis. While heparin-induced thrombocytopenia and clinically relevant osteoporosis seems relatively uncommon, the incidence of major and overall bleeding appears to be comparable between LMWH and VKAs at least for the first 3-6 months of therapy. 6-8 The costs of long-term LMWH administration which exceeds by far that of VKAs 14 as well as the patient's preference should be taken into account when deciding on the optimal long-term VTE prophylaxis.

The optimal anticoagulant prophylaxis in cancer patients with VTE who have completed 6 months of LMWH remains a dilemma. While current guidelines by the American Society of Clinical Oncology and the American College of Chest Physicians advice lifelong LMWH, these recommendations remain based solely on expert consensus in the absence of clinical trial data. A recent worldwide survey has shown that VKAs remain the most commonly used long-term in cancer patients. 15 The aim of this study is to evaluate whether LMWHs are superior to VKAs in the long-term treatment of symptomatic VTE in cancer patients who completed 6 to 12 months of anticoagulant treatment. As stated above, both medicines have been used for over a decade and their side-effects are widely known. In this study, we will only dictate which anticoagulant should be used for long-term treatment, not whether anticoagulant treatment is indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cancer and confirmed pulmonary embolism (PE) or deep vein thrombosis (DVT) of the leg who have been treated for minimally 6 and maximally 12 months with therapeutic doses of anticoagulants, i.e. LMWH or VKA or a new anticoagulant in a trial
2. Written informed consent
3. Indication for long-term anticoagulant therapy (e.g. because of metastasized disease, chemotherapy)

Exclusion Criteria:

1. Legal age limitations (country specific), minimum age at least 18 years
2. Indications for anticoagulant therapy other than DVT or PE
3. Any contraindication listed in the local labeling of LMWH or VKA
4. Childbearing potential without proper contraceptive measures, pregnancy or breastfeeding
5. Life expectancy <3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Symptomatic recurrent VTE, i.e. the composite of recurrent deep venous thrombosis and fatal or non-fatal pulmonary embolism | 6 months
  Primary efficacy outcome

SECONDARY OUTCOMES:
All clinically relevant bleeding (i.e. major bleeding and other clinically relevant non-major bleeding) | 6 months
  safety outcome
all-cause mortality | 6 months
  safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: Pieter W. Kamphuisen, MD, PhD, Principal Investigator — University Medical Center Groningen; Harry R. Buller, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Steering Board Committee, Study Chair — Representatives from participating centers
Locations (14):
- George Washington University, Washington D.C., District of Columbia, United States
- University Health Network, Toronto, Ontario, Canada
- Medical Clinic Dresden University, Dresden, Germany
- Italy (5):
  - Ospedali Riuniti, Bergamo
  - Hospital d'Annunziata, Chieti
  - Ospedaliera di Padova, Padua
  - Arcispedale Santa Maria Nuova (ASMN), Reggio Emilia
  - Ospedale di Circolo, Varese
- Netherlands (6):
  - Flevoziekenhuis, Almere Stad
  - Academic Medical Centre (AMC), Amsterdam
  - Slotervaart Hospital, Amsterdam
  - Reinier de Graaf Groep, Delft
  - Medisch Spectrum Twente, Enschede
  - University Medical Centre Groningen (UMCG), Groningen

REFERENCES:
- [Background] Lee AY, Levine MN, Baker RI, Bowden C, Kakkar AK, Prins M, Rickles FR, Julian JA, Haley S, Kovacs MJ, Gent M; Randomized Comparison of Low-Molecular-Weight Heparin versus Oral Anticoagulant Therapy for the Prevention of Recurrent Venous Thromboembolism in Patients with Cancer (CLOT) Investigators. Low-molecular-weight heparin versus a coumarin for the prevention of recurrent venous thromboembolism in patients with cancer. N Engl J Med. 2003 Jul 10;349(2):146-53. doi: 10.1056/NEJMoa025313. PMID 12853587
- [Background] Meyer G, Marjanovic Z, Valcke J, Lorcerie B, Gruel Y, Solal-Celigny P, Le Maignan C, Extra JM, Cottu P, Farge D. Comparison of low-molecular-weight heparin and warfarin for the secondary prevention of venous thromboembolism in patients with cancer: a randomized controlled study. Arch Intern Med. 2002 Aug 12-26;162(15):1729-35. doi: 10.1001/archinte.162.15.1729. PMID 12153376
- [Background] Lyman GH, Khorana AA, Falanga A, Clarke-Pearson D, Flowers C, Jahanzeb M, Kakkar A, Kuderer NM, Levine MN, Liebman H, Mendelson D, Raskob G, Somerfield MR, Thodiyil P, Trent D, Francis CW; American Society of Clinical Oncology. American Society of Clinical Oncology guideline: recommendations for venous thromboembolism prophylaxis and treatment in patients with cancer. J Clin Oncol. 2007 Dec 1;25(34):5490-505. doi: 10.1200/JCO.2007.14.1283. Epub 2007 Oct 29. PMID 17968019
- [Background] Geerts WH, Bergqvist D, Pineo GF, Heit JA, Samama CM, Lassen MR, Colwell CW. Prevention of venous thromboembolism: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):381S-453S. doi: 10.1378/chest.08-0656. PMID 18574271